CLINICAL TRIAL: NCT01600456
Title: Optimizing PTSD Treatment: PE Versus PE Plus Sertraline
Brief Title: Optimizing Posttraumatic Stress Disorder Treatment: Prolonged Exposure (PE) Versus PE Plus Sertraline
Acronym: OPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University of Washington (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Norah Feeny, Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Optimizing1; R01MH066348-07 (NIH); R01MH066347-07 (NIH)
Record Dates: First submitted 2012-05-11; First posted 2012-05-17 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Antidepressants; Cognitive behavior therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sertraline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Choice: Prolonged exposure (PE) (Active Comparator): Participants randomized to "choice" who choose prolonged exposure (PE).
  Interventions: Behavioral: Prolonged exposure (PE)
- Choice: PE plus sertraline (Active Comparator): Participants randomized to "choice" who choose PE plus sertraline.
  Interventions: Behavioral: Prolonged exposure (PE); Other: PE plus Sertraline
- No choice: Prolonged exposure (PE) (Active Comparator): Participants randomized to "no choice" who are then randomized to PE.
  Interventions: Behavioral: Prolonged exposure (PE)
- No Choice: PE plus sertraline (Active Comparator): Participants randomized to "no choice" who are then randomized to PE plus sertraline.
  Interventions: Behavioral: Prolonged exposure (PE); Other: PE plus Sertraline

INTERVENTIONS:
Behavioral: Prolonged exposure (PE) — PE will include 10 weekly sessions of individual cognitive behavioral therapy.
Other: PE plus Sertraline — PE plus sertraline will include 10 weeks of prolonged exposure therapy plus sertraline. The sertraline dose will be up to 200 mg daily for 10 weeks. There will also be frequent meetings with study psychiatrist. PE will be provided 1x weekly for 10 weeks.
  Other Names: Zoloft
  Arms: Choice: PE plus sertraline; No Choice: PE plus sertraline

SUMMARY:
The specific aims of this study are:

1. To compare the effectiveness of a cognitive behavioral therapy (prolonged exposure, PE) to that of PE and medication (sertraline).
2. To compare the durability of PE gains to that of PE and sertraline at 3, 6, and 9 months post-treatment.
3. To compare those who have chosen their treatment to those who have not in terms of completion of treatment, treatment satisfaction, and short- and long-term effectiveness of the treatment.
4. To examine cost effectiveness of treatment delivery to trauma survivors with PTSD.

DETAILED DESCRIPTION:
Exposure to traumatic events, such as automobile accidents and physical or sexual assault, can cause individuals to develop persistent psychological difficulties such as post-traumatic stress disorder (PTSD). PTSD is an anxiety disorder characterized by avoidance, hyperarousal symptoms, and mental re-experiencing of the traumatic event. PTSD is a serious condition that may cause social and psychological impairment; therefore, safe and effective treatments are needed. Both CBT (cognitive behavior therapy) and antidepressant therapy have been shown to effectively treat PTSD symptoms; however, comparisons of the treatments are limited. This study will compare the short- and long-term effectiveness of prolonged exposure and prolonged exposure plus the antidepressant sertraline.

Participants will either be randomly assigned to prolonged exposure (PE) or PE plus sertraline, or they will be able to choose one of the two treatments,which will be given for 10 weeks, followed by 9 months of follow-up assessments. Participants in the PE group will have 10 weekly sessions of therapy. During the therapy sessions, participants will be encouraged to confront their general fears and the memory of their trauma through repeated storytelling. Participants will also be encouraged to practice the techniques learned in therapy in everyday life. Participants in the PE plus sertraline group receive the same treatment as the PE group plus they will take sertraline daily for 10 weeks. These participants will be seen regularly by a psychiatrist who will offer general encouragement and support, monitor response to medication, and record any side effects participants may be experiencing. The medication may be adjusted according to a dosing schedule and based on the study doctor's judgment. At the end of 10 weeks, participants in the PE plus sertraline group will have the choice of either tapering the medication gradually to minimize the chance of withdrawal symptoms or staying on the medication for up to 9 months. Participants who do not respond to their assigned or chosen treatment will be offered booster sessions or the other treatment for 10 weeks. Self-report scales and questionnaires will be used to assess participants' PTSD symptoms, depression, anxiety, and social functioning. These assessments will occur at 3, 6, and 9 months after the study treatment period.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV (Diagnostic & Statistical Manual of Mental Disorders) diagnosis of PTSD (with severity threshold)
* Experienced traumatic event at least 12 weeks prior to study entry
* Willingness to discontinue current CBT or antidepressant treatment if needed

Exclusion Criteria:

* Current diagnosis of schizophrenia or delusional disorder
* Medically unstable bipolar disorder, depression with psychotic features, or depression requiring immediate psychiatric treatment
* No clear trauma memory or trauma before age 3
* Current diagnosis of alcohol or substance dependence within 3 months prior to study entry
* Ongoing intimate relationship with the perpetrator of the traumatic event
* History of nonresponse to adequate trial of either CBT or sertraline
* Medical contraindication for sertraline
* Current high dose use of benzodiazepines
* Pregnant or sexually active female without adequate birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Posttraumatic stress disorder (PTSD) Symptoms | Measured up to 9 months.
  Interview measure to assess PTSD symptoms.

SECONDARY OUTCOMES:
Depression symptoms | Measured up to 9 months.
  Clinical assessment of depression symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Norah C Feeny, PhD, Principal Investigator — Case Western Reserve University; Lori A Zoellner, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Psychological Sciences Department Case Western Reserve University, Cleveland, Ohio
  - Psychology Department of University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Rosencrans PL, Walker RSW, Coyne AE, Baier AL, Klein AB, Shekhtman K, Bowling AR, Feeny NC, Zoellner LA. Reciprocal relationships between posttraumatic stress disorder symptoms and positive and negative affect in evidence-based treatments for posttraumatic stress disorder. J Consult Clin Psychol. 2024 Sep;92(9):630-640. doi: 10.1037/ccp0000898. PMID 39418460
- [Derived] Coyne AE, Mattson E, Bagley JM, Klein AB, Shekhtman K, Payat S, Levine DS, Feeny NC, Zoellner LA. Within-patient association between emotion regulation and outcome in prolonged exposure for posttraumatic stress disorder. J Consult Clin Psychol. 2024 Sep;92(9):582-593. doi: 10.1037/ccp0000837. Epub 2023 Nov 16. PMID 37971811
- [Derived] Rosencrans PL, Zoellner LA, Feeny NC. A network approach to posttraumatic stress disorder: Comparing interview and self-report networks. Psychol Trauma. 2024 Feb;16(2):340-346. doi: 10.1037/tra0001151. Epub 2021 Oct 21. PMID 34672659
- See also: Optimizing PTSD Treatment's Homepage — http://www.ptsdoptions.com